CLINICAL TRIAL: NCT02858947
Title: Three-Year Clinical Evaluation of Class II Posterior Composite Restorations Placed With Different Techniques and Flowable Composite Linings in Endodontically Treated Teeth
Brief Title: Three-Year Clinical Evaluation of Class II Posterior Composite Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Dr Emel Karaman, Assistant professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMU-TAEK 2011/482
Record Dates: First submitted 2016-07-26; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Dental Caries
Keywords: composite resin; bulk-fill; teeth endodontically-treated
MeSH Terms: conditions — Dental Caries; Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aelite Flo (Active Comparator): Microhybrid flowable composite
  Interventions: Procedure: Aelite Flo
- x-tra base (Active Comparator): Bulk-fill flowable composite
  Interventions: Procedure: x-tra base

INTERVENTIONS:
Procedure: Aelite Flo — Microhybrid flowable composite
  Other Names: 1000006652
  Arms: Aelite Flo
Procedure: x-tra base — Bulk-fill flowable composite
  Other Names: 1145403
  Arms: x-tra base

SUMMARY:
The aim of this study was to investigate the clinical effectiveness of direct resin composite restorations placed with different placement techniques (incremental or bulk) and with different flowable linings (conventional or bulk-fill flowable) used in open-sandwich technique, in endodontically treated Class II cavities (mesio-occlusal or disto-occlusal), in a randomized controlled comparison.

DETAILED DESCRIPTION:
Forty-seven pairs Class II (mesio-occlusal or disto-occlusal) composite restorations were placed in 37 patients. In all cavities, Adper Single Bond 2 was used. In one of the cavities of each pair, a conventional flowable composite, Aelite Flo, was applied in approximately 2mm thick, and the remaining cavity was restored incrementally with GrandioSO. In the second cavity, a bulk-fill flowable composite, x-tra base, was applied in approximately 4 mm thick in bulk increments and the remaining 2mm occlusal part of the cavity was restored with GrandioSO. All cavities were restored with open-sandwich technique by the same operator. At baseline and after 6-month, 1-, 2- and 3-year follow-up visits, restorations were evaluated by Modified USPHS criteria.

ELIGIBILITY:
Inclusion Criteria:

* Permanent premolars and molars without any restorations were included in the study. Every tooth included in the study had neighboring teeth and were in occlusion to antagonistic teeth.

Exclusion Criteria:

* Patients were excluded who needed indirect restorations due to significant loss of tooth structure, known allergies to product ingredients, had poor oral hygiene and a history of bruxism.

Ages: 19 Years to 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2011-03; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance evaluation of different composite resin restorations with USPHS criteria | three years
  Every year in three years period

IPD SHARING:
Plan to Share IPD: No